CLINICAL TRIAL: NCT07197892
Title: Conversational AI Platform for Early Pregnancy Care City-wide Recruitment: A Feasibility Study
Acronym: CIRCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 859274
Record Dates: First submitted 2025-09-26; First posted 2025-09-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Early Pregnancy
Keywords: Early pregnancy loss; Miscarriage; Prenatal care; Abortion
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CIRCA Texting Platform (Experimental): CIRCA is a two-way texting platform that uses artificial intelligence to match patient texts to clinician-vetted responses and send educational content.
  Interventions: Other: CIRCA Texting Platform

INTERVENTIONS:
Other: CIRCA Texting Platform — Two-way texting platform that uses artificial intelligence to match patient texts to clinician-vetted responses and send educational content

SUMMARY:
This study seeks to determine pregnant patients in the Philadelphia area can be recruited to a conversational AI texting platform. The trial will be considered feasible if recruitment goals are met in proportion to delivery volume at the hospital.

DETAILED DESCRIPTION:
The investigators developed a conversational AI platform to improve periconception care (CIRCA) to engage individuals in their healthcare decision making, reduce barriers to care, and ultimately reduce widespread inequities in reproductive and maternal health.

CIRCA was developed to enable care from positive pregnancy test onward. After a positive test, patients scan a QR code to onboard via SMS to the program. A positive pregnancy test is confirmed, and an estimated gestational duration is calculated from last menstrual period, if known. If unknown, the patient is directed to schedule a visit at a nearby early pregnancy assessment center where they can receive routine testing and counseling to confirm the pregnancy and its gestational duration. They are then able to receive triage and scheduled educational content.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Access to a working mobile phone
* Ability to read English
* Pregnant with a gestational age less than 12 weeks, 6 days by last menstrual period or by ultrasound, or per patient self-report

Exclusion Criteria: N/A

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2637 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of citywide recruitment of pregnant patients in Philadelphia. | 12 months
  Proportion of pregnant patients in Philadelphia who sign up to use CIRCA texting platform

SECONDARY OUTCOMES:
Platform engagement | Between platform enrollment up until 12 weeks, 6 days gestation
  Percentage of surveys completed by participant
Platform acceptability | To be completed at 1 week of use and at final study survey (up to 12 weeks 6 days gestation)
  Net promoter score (Range 0-10, with a higher score indicating a better rating)
Birth outcome | From platform enrollment up until the event of a live birth or other pregnancy outcome.
  Early pregnancy loss, ectopic pregnancy, abortion, severe maternal morbidity, preterm birth
Emergency Department Utilization | From platform enrollment until 12 weeks, 6 days gestation.
  Emergency Department visits

CONTACTS AND LOCATIONS:
Overall Officials: Alice Abernathy, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No